CLINICAL TRIAL: NCT02433600
Title: The Effect of Feeding Infant Formula With Enriched Protein Fractions
Brief Title: The Effect of Feeding Infant Formula With Enriched Protein Fractions in the US
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to lack of enrollment
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 6035
Record Dates: First submitted 2015-04-27; First posted 2015-05-05 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Declarative Memory

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cow's milk-based infant formula (Active Comparator)
  Interventions: Other: Cow's milk-based infant formula
- Cow milk-based infant formula with enriched protein fractions (Experimental)
  Interventions: Other: Cow milk-based infant formula with enriched protein fractions

INTERVENTIONS:
Other: Cow's milk-based infant formula
  Arms: Cow's milk-based infant formula
Other: Cow milk-based infant formula with enriched protein fractions
  Arms: Cow milk-based infant formula with enriched protein fractions

SUMMARY:
This study is intended to measure declarative or stored memory and behavior between infants who consume one of two infant formulas through approximately one year of age.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, 0-90 days of age at randomization
* Term infant with birth weight of a minimum of 2500 grams
* Receiving at least 75% of the recommended caloric intake from cow's milk-based infant formula
* Parent or legally authorized representative attending study visits reads, understands, and speaks English
* Signed Informed Consent and Protected Health Information authorization

Exclusion Criteria:

* History of underlying metabolic or chronic disease, congenital malformation, or immunocompromised
* Feeding difficulties or formula intolerance
* Infant born small for gestational age
* Infant born from a mother who was diabetic at childbirth
* History of seizures or neurological disorders or infant with known head/brain disease/injury

Max Age: 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Sequence Recall using 3-dimensional props | 365 days of age

SECONDARY OUTCOMES:
Electroencephalogram response to stimuli | 180 days of age
Sequence Recall using 3-dimensional props | 300 days of age
Infant Behavior Questionnaire Revised, Short | 240 days of age
MacArthur-Bates Communication Development Inventory | 365 days of age
Bayley Scales of Infant and Toddler Development, Third Edition | 365 days of age
Achieved Weight | 52 weeks
Achieved Length | 52 weeks
Achieved Head Circumference | 52 weeks
Formula Intake | 52 weeks
Medically-confirmed Adverse Events | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lynn Berseth, MD, Study Director — Mead Johnson Nutrition
Locations (1):
- University or North Carolina Nutrition Research Instutite, Kannapolis, North Carolina, United States

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831